CLINICAL TRIAL: NCT04055168
Title: A Phase I Randomized Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD6615 After Single Dosing to Healthy Subjects
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD6615 in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: It was decided to not run the Japanese cohorts in the study.
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D7991C00001
Record Dates: First submitted 2019-07-15; First posted 2019-08-13 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Dyslipidemia
Keywords: Dyslipidemia; Single Ascending Dose; Safety; Tolerability
MeSH Terms: conditions — Dyslipidemias | interventions — Drug Evaluation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 - Part 1 (Experimental): On Day 1, randomized subjects (healthy non-Asian subjects) will receive dose 1 of AZD6615 (6 subjects) or matching placebo (2 subjects).
  Interventions: Drug: AZD6615; Drug: Placebo
- Cohort 2 - Part 1 (Experimental): On Day 1, randomized subjects (healthy non-Asian subjects) will receive dose 2 of AZD6615 (6 subjects) or matching placebo (2 subjects).
  Interventions: Drug: AZD6615; Drug: Placebo
- Cohort 3 - Part 1 (Experimental): On Day 1, randomized subjects (healthy non-Asian subjects) will receive dose 3 of AZD6615 (6 subjects) or matching placebo (2 subjects).
  Interventions: Drug: AZD6615; Drug: Placebo
- Cohort 1 - Part 2 (Experimental): On Day 1, randomized subjects (healthy Japanese subjects) will receive dose 1 of AZD6615 (6 subjects) or matching placebo (2 subjects).
  Interventions: Drug: AZD6615; Drug: Placebo
- Cohort 2 - Part 2 (Experimental): On Day 1, randomized subjects (healthy Japanese subjects) will receive dose 2 of AZD6615 (6 subjects) or matching placebo (2 subjects).
  Interventions: Drug: AZD6615; Drug: Placebo

INTERVENTIONS:
Drug: AZD6615 — AZD6615 (dose 1, dose 2, or dose 3) will be administered as a single dose to the randomized subjects.
  Other Names: Study drug
Drug: Placebo — Placebo (dose 1, dose 2, or dose 3) will be administered as a single dose to the randomized subjects.
  Other Names: Control

SUMMARY:
This study will be a randomized, single-blind, placebo-controlled, single-ascending dose (SAD), sequential group study. It is a SAD study in healthy Non-Asian subjects (Part 1) and healthy Japanese subjects (Part 2) to assess the safety and tolerability of AZD6615 and to characterize the pharmacokinetics (PK) of AZD6615.

DETAILED DESCRIPTION:
This study part is planned to consist of 3 cohorts of Non-Asian subjects (Part 1) and 2 cohorts of Japanese subjects (Part 2). Part 2 will be initiated no earlier than after completion of the last Safety Review Committee (SRC) review in Part 1. Healthy male and/or female subjects aged 20 to 60 years will be included in both Parts 1 and 2 of the study. Female subjects must be of non-childbearing potential. Study Part 1 is planned to be conducted in 24 subjects but may be conducted in up to 40 subjects. Study Part 2 is planned to be conducted in 16 subjects but may be conducted in up to 32 subjects.

Within each cohort of Parts 1 and 2, 6 subjects will be randomized to receive AZD6615 and 2 subjects will be randomized to receive placebo. Dosing and food intake should be supervised and documented by study staff when subjects are in the clinic.

The study will comprise of:

* A Screening Period of maximum 28 days.
* A Dosing Session during which subjects will be resident at the Clinical Unit from the day before IMP administration (Day -1) until at least 78 hours after Investigational medicinal product (IMP) administration; discharged on Day 4.
* A Follow-Up Period of 12 weeks that will consist of 6 Follow-Up Visits, for which the subjects will return to the Clinical Unit at 2, 4, 6, 8, 10, and 12 weeks post-dose.

Within each cohort, site personnel remain blinded until the SRC meeting.

Following review of the data, the SRC may also decide to adjust the following for subsequent cohorts:

* The time window between the sentinel dose group and the main dose group in Part 1.
* The length of the stay at the study site, the timing and number of assessments and/or samples.
* The length of the follow-up period.
* The length of the data collection period for the SRC review.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit, must not be lactating and must be of non-child-bearing potential.
3. Provision of signed, written and dated informed consent for optional genetic research.

4: In Part 1: Healthy male and/or female Non-Asian subjects aged 20 - 60 years (inclusive at Screening Visit) with suitable veins for cannulation or repeated venipuncture. In Part 2: Healthy male and/or female Japanese subjects aged 20 - 60 years (inclusive at Screening Visit) with suitable veins for cannulation or repeated venipuncture.

5. Have a body mass index between 18 and 30 kg/m^2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive at the Screening Visit and Day -1.

6. Males should avoid fathering a child by either true abstinence or a highly effective contraception form of birth control during the study.

Exclusion Criteria:

1. History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
3. Subjects with known autoimmune disease or on treatment with immune-modulatory drugs.
4. Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the administration of investigational medicinal product.
5. Any laboratory values with the following deviations at the Screening Visit and/or Day -1, test may be repeated once for each visit at the discretion of the Investigator if out of range: (Alanine aminotransferase > upper limit of normal [ULN], Aspartate aminotransferase > ULN, Creatinine > ULN, White blood cell count < 3.5 x 10^9/L, Hb < lower limit of normal [LLN], Platelet count <LLN).
6. Any positive result on Screening for serum hepatitis B surface antigen, hepatitis C antibody and human immunodeficiency virus.
7. Abnormal vital signs, any clinically important abnormalities in rhythm, conduction or morphology of the resting ECG and any clinically important abnormalities in the 12-Lead ECG as considered by the Investigator, that may interfere with the interpretation of QTc interval changes.
8. Known or suspected history of drug abuse, current smoker or those who have smoked or used nicotine products within the previous 3 months before the Screening Visit.
9. History of alcohol abuse and/or severe allergy/hypersensitivity.
10. Previous bone marrow transplant.
11. Males who are unwilling to use an acceptable method of birth control during the entire study period.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs) and serious adverse events (SAEs) | From screening to 12 weeks of follow-up
  To assess the safety and tolerability of AZD6615 following the administration of SAD

SECONDARY OUTCOMES:
Plasma PK analysis: Maximum observed concentration (Cmax) | Days 1 to 4: Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose
  To characterize the PK of AZD6615 after single dosing
Plasma PK analysis: Time to reach maximum observed concentration (tmax) | Days 1 to 4: Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose
  To characterize the PK of AZD6615 after single dosing
Plasma PK analysis: Terminal half-life (t½λz) | Days 1 to 4: Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose
  To characterize the PK of AZD6615 after single dosing
Plama PK analysis: Terminal elimination rate constant (λz) | Days 1 to 4: Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose
  To characterize the PK of AZD6615 after single dosing
Plasma PK analysis: Area under the plasma concentration-curve from time zero to the time of last quantifiable analyte concentration (AUClast) | Days 1 to 4: Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose
  To characterize the PK of AZD6615 after single dosing
Plasma PK analysis: Area under the plasma concentration-time curve from time zero to 24 hours after dosing (AUC0-24) | Days 1 to 4: Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose
  To characterize the PK of AZD6615 after single dosing
Plasma PK analysis: Area under the concentration-time curve from time zero extrapolated to infinity (AUC) | Days 1 to 4: Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose
  To characterize the PK of AZD6615 after single dosing
Plasma PK analysis: Apparent volume of distribution (Vz/F) | Days 1 to 4: Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose
  To characterize the PK of AZD6615 after single dosing
Plasma PK analysis: Apparent total body clearance (CL/F) | Days 1 to 4: Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose
  To characterize the PK of AZD6615 after single dosing
Plasma PK analysis: Area under the plasma concentration-time curve from time zero extrapolated to infinity divided by the dose administered (AUC/D) | Days 1 to 4: Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose
  To characterize the PK of AZD6615 after single dosing
Plasma PK analysis: Area under the plasma concentration-time curve from time zero to 24 hours after dosing divided by the dose administered (AUC0-24/D) | Days 1 to 4: Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose
  To characterize the PK of AZD6615 after single dosing
Plasma PK analysis: Area under the plasma concentration-time curve from time zero to time of last quantifiable analyte concentration divided by the dose administered (AUClast/D) | Days 1 to 4: Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose
  To characterize the PK of AZD6615 after single dosing
Plama PK analysis: Mean Residence Time from time 0 to infinity (MRT) | Days 1 to 4: Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose
  To characterize the PK of AZD6615 after single dosing
Plasma PK analysis: Observed maximum concentration divided by the dose administered (Cmax/D) | Days 1 to 4: Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose
  To characterize the PK of AZD6615 after single dosing
PD analysis: Levels of dyslipidemia related biomarkers | At screening, on Days -1, Days 1 to 4 (Pre-dose and at 24, 48 and 72 hours post-dose), Weeks 2 to 10 (at 2, 4, 6 and 8 weeks post-dose) and on Week 12 post-dose
  This study will also investigate the PD of AZD6615 by investigating the effect of AZD6615 on levels of dyslipidemia related biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: David Han, MD, Principal Investigator — California Clinical Trials Medical Group
Locations (2):
- United States (2):
  - Research Site, Glendale, California
  - Research Site, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Makhmudova U, Steinhagen-Thiessen E, Volpe M, Landmesser U. Advances in nucleic acid-targeted therapies for cardiovascular disease prevention. Cardiovasc Res. 2024 Sep 2;120(10):1107-1125. doi: 10.1093/cvr/cvae136. PMID 38970537